CLINICAL TRIAL: NCT04300179
Title: Ewing Sarcoma Family of Tumors (ESFT): A 15-year Experience From a Tertiary Care Cancer Center in Upper Egypt
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Morsy, MD, Lecturer of Pediatric Oncology, Assiut University
Other Study IDs: ESFT_Upp_Egypt
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Soft Tissue Neoplasms; Bone Neoplasms; Neoplasms
Keywords: Ewing's sarcoma (ES); Peripheral primitive neuroectodermal tumor (PNET)
MeSH Terms: conditions — Soft Tissue Neoplasms; Bone Neoplasms; Neoplasms; Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify demographic & disease characteristics in pediatric oncology patients diagnosed with Ewing Sarcoma Family of Tumors (ESFT) & treatment outcomes in these patients.

DETAILED DESCRIPTION:
Ewing sarcoma (ES) and peripheral primitive neuroectodermal tumor (PNET), Both entities that currently comprise the same spectrum of neoplastic diseases known as the Ewing sarcoma family of tumors (EFT), were originally described as distinct clinicopathologic entities. Primitive neuroectodermal tumors (PNETs) first described in 1918 by Stout as a malignant tumor arising from major nerve. Later, in 1921, ES was described as an undifferentiated tumor involving the diaphysis of long bones. It was also reported to arise in soft tissue (extraosseous ES). EFT is aggressive malignant small round cell tumors of bone and soft-tissue that predominantly affecting children and young adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose age less than 19 years. Patients diagnosed with Ewing Sarcoma Family of Tumors (ESFT).

Exclusion Criteria:

* Patients whose age more than 19 years. Patients diagnosed with other bone & soft tissue neoplasms.

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cancer patients, those diagnosed with Ewing Sarcoma Family of Tumors (ESFT), in the period from 2000 January till 2015 December, and received treatment at the pediatric oncology department, their medical records will be retrospectively reviewed for data collection.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-12-16 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of treatment initiation until the date of death from any cause or patients censored at last follow up, whichever came first, assessed up to 60 months
  Participants will be retrospectively followed forward in time from the date of initiation of treatment till death from any cause, an expected average of 5 years
Event Free Survival (EFS) | From date of treatment initiation until the date of event from any cause or patients censored at last follow up, whichever came first, assessed up to 60 months
  Participants will be retrospectively followed forward in time from the date of initiation of treatment till occurrence of an event from any cause (tumor progression, relapse) or death, an expected average of 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt